CLINICAL TRIAL: NCT02207933
Title: Effect of Anterioposterior Weight Shifting Training With Visual Biofeedback in Patients With Step Length Asymmetry After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4-2013-0270
Record Dates: First submitted 2014-07-31; First posted 2014-08-04 (Estimated); Last update posted 2019-03-27 (Actual); Status verified 2014-12

CONDITIONS: Stroke; Hemiplegic Gait
Keywords: anterioposterior; weight; shifting; training; patient
MeSH Terms: conditions — Stroke; Gait Disorders, Neurologic; Body Weight

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- AP shifting group (Experimental)
  Interventions: Procedure: AP shifting training
- gait training group (Active Comparator)
  Interventions: Procedure: Gait training

INTERVENTIONS:
Procedure: AP shifting training — AP shifting training in addition to gait training 3 times a week for 6 weeks
  Arms: AP shifting group
Procedure: Gait training — Gait training only for 3 times a week for 6 weeks.
  Arms: gait training group

SUMMARY:
To investigate the effect of anteroposterior weight shifting training with visual biofeedback on step length asymmetry. Reduced speed and asymmetry of stepping is a specific characteristic of hemiplegic gait. Asymmetry of stepping is characterized by shorter step length of the unaffected limb compared to the affected limb. Causes of this phenomenon are difficulty in weight bearing at the affected limb, weak propulsive force of the affected limb, and decreased strength of hip extensors. To correct these factors. we have developed an anteroposterior weight shifting training system with visual feedback and studied its effects.

ELIGIBILITY:
Inclusion Criteria:

1. Independent standing
2. Ability to walk 10m without manual assistance
3. Asymmetric ratio of step length > 1.1
4. No severe perceptual, cognitive or cardiovascular impairments that could affect walking

Exclusion Criteria:

1. Quadriplegia or double hemiplegia
2. Orthopedic or neurologic conditions in addition to the stroke
3. Had more than 1 cerebrovascular accident

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2013-06; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
change of step Length Asymmetric Ratio | baseline, 3 weeks, 6 weeks, 12 weeks
  paretic step length/non paretic step length

SECONDARY OUTCOMES:
change of Step Length Asymmetric Index | baseline, 3 weeks, 6 weeks, 12 weeks
  paretic step length-non paretic step length/0.5[paretic step length +non paretic step length

CONTACTS AND LOCATIONS:
Overall Officials: Deog Young Kim, MD, PhD, Principal Investigator — Severance Hospital
Locations (1):
- Severance hospital, Seoul, South Korea